CLINICAL TRIAL: NCT05636787
Title: A Randomized Phase II Trial Comparing Treosulfan and Melphalan With Melphalan Alone as Conditioning Regimen for Autologous Stem Cell Transplantation (ASCT) in Myeloma Patients (TreoMel Trial)
Brief Title: Clinical Trial Investigating the Chemotherapeutic Compound Treosulfan (Trecondi® Ideogen) in Myeloma Patients
Acronym: TreoMel
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TreoMel Trial
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Melphalan; Treosulfan
MeSH Terms: conditions — Multiple Myeloma | interventions — treosulfan; Melphalan

STUDY DESIGN:
Intervention Model Description: Randomized prospective non-blinded clinical phase II trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm B - TreoMel (Experimental): Chemotherapy regime consisting of treosulfan on three days at 14 g/m2 followed by 200 mg/m2 melphalan given on two days at 100 mg/m2.
  Interventions: Drug: Treosulfan; Drug: Melphalan
- Arm A - Mel (Active Comparator): Chemotherapy regime consisting of 200 mg/m2 melphalan, split into two days à 100 mg/m2.
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Treosulfan — Efficacy of standard treatment melphalan will be compared to the combination melphalan with treosulfan
  Arms: Arm B - TreoMel
Drug: Melphalan — Efficacy of standard treatment melphalan will be compared to the combination melphalan with treosulfan

SUMMARY:
Clinical trial investigating the chemotherapeutic compound treosulfan (Trecondi® Ideogen) in myeloma patients.

DETAILED DESCRIPTION:
Background and rationale:

Due to demographic changes, multiple myeloma with its preferential manifestation in the elderly population exerts increasing incidence worldwide. Since decades, autologous stem cell transplantation (ASCT) after high-dose chemotherapy (HDCT) with melphalan is the standard first-line consolidation option for patients with multiple myeloma considered fit for this approach. Nevertheless, subsequent relapse despite this intensive treatment is inevitable in most myeloma patients, emphasizing the unmet clinical need for improved conditioning strategies to further enhance the effect of HDCT treatment.

The Inselspital in Bern represents one of the largest European centers for autologous stem cell transplantation (ASCT) in myeloma, lymphoma and leukemia patients, and it is the largest center in Switzerland for ASCT, with more than 150 ASCT performed annually. In parallel, the transplant team at the Inselspital has a dedicated history of clinical trials aiming to further improve tolerance and efficacy of HDCT with ASCT.

In a previous randomized phase 2 study performed at the department of medical oncology of the Inselspital, the combination of the cytotoxic compound bendamustin in addition to the standard melphalan dose as a novel HDCT regimen before autologous transplantation in 120 myeloma patients has been explored and established. This approach was successful in terms of increased anti-myeloma efficacy, but the nephrotoxicity of high-dose bendamustin was relevant in a significant subset of patients. This fact, ultimately, led to the propose of a novel approach.

The present study aims to combine high-dose melphalan (Melphalan Ideogen) with treosulfan (Trecondi® Ideogen), a well established bifunctional alkylating agent. Treosulfan has a favorable toxicity profile, and it is used in patients with acute leukemias in the allogeneic transplant setting as a standard approach in an increasing number of centers. However, no study so far evaluated treosulfan combined with melphalan as high-dose chemotherapy in patients with multiple myeloma. Consequently, this approach is unique and novel in patients with multiple myeloma in the autologous transplant setting.

Compared to the closely related (and more known) compound busulfan, treosulfan compares favorably in terms of decreased neurotoxicity (for busulfan, antiepileptic prophylaxis is necessary), and it does not cause irreversible hair loss, which is often observed after busulfan treatment. The team at the Inselspital performed a pilot study in 25 patients with relapsed myeloma undergoing second-line HDCT/ASCT therapy. Treosulfan (14 mg/m2 i.v. at days -4, -3, and -2) combined with standard dose melphalan (day -1) had promising anti-myeloma activity and was well tolerated as expected from the previous studies. Standardized measurement of treosulfan serum levels by mass spectrometry (Metabolomics, University Institute of Clinical Chemistry, Inselspital Bern) in these patients demonstrated consistent pharmacokinetic profiles with peak levels within the therapeutic range and with low interindividual differences. Consequently, no modifications of the treosulfan dosage were needed during these initial experiences. With the clinical trial outlined in this protocol, the study team aim to gain insights into the use of treosulfan as part of the high-dose chemotherapy regimen before ASCT in myeloma patients. The study will be performed as an open-label, randomized phase 2 study, involving multiple recruiting regional Swiss centers, with all high-dose treatments being performed at the University Hospital Inselspital Bern. Patients will first undergo standardized induction therapy (e.g. VRD regimen, with or without Daratumumab), followed by a 1:1 randomization to two treatment arms:

Arm B, the experimental ("TreoMel") arm, combines treosulfan at three days at 14 g/m2 followed by 200 mg/m2 melphalan given on two days at 100 mg/m2. Arm A, the standard arm, comprises standard 200 mg/m2 melphalan ("Mel"), split into two days à 100 mg/m2.

The stem cell transplantation is identical in both arms, as is the post-transplant management.

In patients with reduced renal function (creatinine clearance <50 mL/min and ≥ 35 ml/min), the melphalan total dose will be lowered to 140 mg/m2, split into two doses at 70 mg/m2. Treosulfan will be administered in a dosage of 14 mg/m2 i.v. on days -5, -4, and -3 in Arm A ("TreoMel"). The autologous cells will be transfused on day 0.

Patients will be stratified 1) according to the myeloma remission status as assessed based on the last available remission status: complete (CR) and very good partial remission (VGPR) versus partial remission (PR), minimal remission (MR), no change (NC) and progressive disease (PD); and 2) according to renal function: Renal function: creatinine clearance ≥ 50 ml/min versus < 50 ml/min.

Based on a previous cohort of 122 myeloma patients at the Inselspital (2010-2013), a CR1 rate in the standard (Mel) arm of 50% is anticipate.

The primary endpoint is to show an improvement of the CR rate after ASCT (before initiation of maintenance treatment) in the standard arm A using melphalan only ("Mel") from 50% to 65% in the experimental arm B combining treosulfan and melphalan ("TreoMel").

Therefore, the study is considered successful if the experimental treosulfan/melphalan arm is superior by 15% points. With a statistical power of 80% and one-tailed significance level of 5%, 60 patients are required for cohorts A and B each. Thus, the total number of patients for the trial needed amounts to 120 patients. As the yearly number of myeloma patients undergoing HDCT/ASCT therapy at the Inselspital Bern is close to 80 patients, the recruitment of a sufficient number of patients in the planned study duration of 36 months appears feasible.

Patients can be included with a diagnosis of multiple myeloma after standard first-line induction therapy, commonly being the VRD regimen with or without additional daratumumab. In the case of refractory myeloma, one or several additional alternative induction regimens can be applied before the study treatment. Further preconditions are clinical fitness for HDCT/ASCT and age of at least 18 years, ECOG less than 3, and creatinine clearance of at least 35 mL/min or more (for additional incl./excl. criteria see the entire protocol).

The measurement of the endpoints of the study will be as follows: Primary endpoint is the complete remission (CR) rate after ASCT (before initiation of maintenance treatment) following measurement of myeloma parameters in the peripheral blood including M-gradient, quantitative immunoglobulins, kappa/lambda light chain ratio, and immunofixation. Secondary endpoints are: time to neutrophil and thrombocyte engraftment, progression-free and overall survival, toxicities, infectious complications, hospitalization duration, minimal residual disease (MRD) load determined by next-generation immunophenotyping. Treosulfan serum levels will be assessed by pharmacokinetic drug monitoring based on mass spectrometry. Bone marrow punction for defining the response will be performed in all patients after neutrophil engraftment before hospital discharge around 15 days after ASCT. Bone marrow analyses comprise cytomorphology, histopathology, and flow cytometry at a sensitivity level of 10(-5) for MRD assessment.

The trial will be performed at the Department of Oncology at the Inselspital, University Hospital Bern. The CTU of the University of Bern will perform the on-site monitoring of the study.

ELIGIBILITY:
Inclusion criteria:

1. Eligible are myeloma patients after standard first-line induction treatment. Additional induction regimens in refractory myeloma patients are allowed.
2. Patients must be considered fit for subsequent consolidation with high-dose chemotherapy with autologous stem cell transplantation.
3. Patients must be aged 18-75 years.
4. Patients must have an ECOG <3.
5. Patients must have a creatinine clearance ≥35 ml/min.
6. Patients must have an LVEF ≥40% within three months prior to start of study HDCT.
7. Patients must have given voluntary written informed consent.

Exclusion criteria:

1. Patients with an uncontrolled acute infection.
2. Patients with a transplantation comorbidity index (HCTCI) > 6 points.
3. Patients with concurrent active malignant disease with the exception of basalioma/spinalioma of the skin or early-stage cervix carcinoma, or early-stage prostate cancer. Previous treatment for other malignancies (not listed above) must have been terminated at least 6 months before registration and no evidence of active disease may be documented since then.
4. Patients with major coagulopathy or bleeding disorder.
5. Patients with other medical conditions that could potentially interfere with the completion of treatment according to this protocol or that would impair tolerance to therapy or prolong hematological recovery.
6. Lack of patient cooperation to allow study treatment as outlined in this protocol.
7. Known pregnancy or lactating female patients. The pregnancy test could be omitted from the screening visit and postponed to the study treatment if indicated (a pregnancy test in female patients of child-bearing potential is not mandatory since patients are already under induction chemotherapy or mobilization chemotherapy, and pregnancy was excluded before starting induction chemotherapy; if, however, a pregnancy test is clinically indicated, it can be done either during screening or before the start of study treatment).

   Patient not willing to implement adequate contraceptive measures (hormonal treatment p.o. or i.m., intra-uterine surgical devices, or latex condoms) to avoid pregnancy during study treatment and for 12 additional months.
8. Use of any anti-cancer investigational agents within 14 days prior to the expected start of trial treatment.
9. Contraindications and hypersensitivity to any of the active chemotherapy compounds.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Complete Remission (CR) Rate | 15 days after ASCT
  Number of patients experiencing CR ( Myeloma assessment (serum free light chain ratio, M-gradient, IgG, IgA, IgM), Flow cytometry MRD, FISH analysis (plasma), Bone marrow (aspirate and biopsy) is performed only in patients fulfilling the criteria for CR. Bone marrow should be assessed at the end of the ASCT hospitalization)

SECONDARY OUTCOMES:
Adverse Events | 15 days after ASCT
  Number of patient experiencing toxicity (Assessment of CTCAE V5.0 highest toxicity score observed for toxicities of at least grade 3)
Infectious complications | 15 days after ASCT
  Number of patients experiencing infectious complications
Engraftment and hematologic recovery | 15 days after ASCT
  Number of days until neutrophils recovery 0.5 G/L (from day -5) and platelet recovery 20 G/L
Renal toxicity | 15 days after ASCT
  Number of patients experiencing renal toxicity (>1.5-3.0 x baseline)
Overall survival | 5 years
  Days from ASCT until death of any cause or date of last follow-up
Progression free survival | 5 years
  Days from ASCT until first recurrence of myeloma or date of last follow-up
Hospitalisation duration | 30 days
  Days staying in hospital
Minimal residual disease (MDR) | 30 days
  Assessed by flow cytometry from bone marrow samples
Pharmacodynamics of Treosulfan | Day -4
  Assessed by mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pabst, Prof Dr. med, Study Chair — Department for Medical Oncology; University Hospital/Inselspital
Locations (1):
- Departement of Medical Oncology, University Hospital Berne, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes